CLINICAL TRIAL: NCT02881723
Title: Obstructive Sleep Apnea Syndrome After Oropharyngeal Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-25; 2012-A00863-40 (Other: ANSM)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea Syndrome; Oropharyngeal Cancer
MeSH Terms: conditions — Sleep Apnea, Obstructive; Oropharyngeal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment for oropharyngeal cancer by surgery (Experimental): Disease-free patients treated for locally advanced oropharyngeal cancer for over 12 months by surgery
  Interventions: Procedure: Surgery
- Treatment for oropharyngeal cancer by radio-chemotherapy (Experimental): Disease-free patients treated for locally advanced oropharyngeal cancer for over 12 months by radio-chemotherapy
  Interventions: Radiation: Radio- chemotherapy

INTERVENTIONS:
Procedure: Surgery
  Arms: Treatment for oropharyngeal cancer by surgery
Radiation: Radio- chemotherapy
  Arms: Treatment for oropharyngeal cancer by radio-chemotherapy

SUMMARY:
The level of knowledge about the consequences of oropharyngeal cancer treatment on sleep quality remains poor. Because of a high level of risk of developing an Obstructive Sleep Apnea Syndrome (OSAS), an accurate evaluation of the prevalence, of the risk factors and of the impact on quality of life is important in order to propose preventive and therapeutic solutions to these patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) remains poorly documented in head and neck cancer cancer population, who have a higher risk than the general population. OSAS is a risk factor for quality of life impairment and cardiovascular morbidity and mortality.

This study proposes to carry out an OSAS prevalence study among a locally advanced head and neck cancer population, already treated and to compare the consequences of current therapeutic options in sleep quality.The primary research objective will be a prevalence determination in a locally advanced stages treated population of oropharyngeal cancer. Secondary objectives will be the comparison of the prevalence between the surgical group and the radio-chemotherapy group, the research of predictive factors of presenting an OSAS and the precision of the impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old, male or female;
* Patient treated for a first oropharyngeal cancer located in upper airways (velum, side walls, back wall, base of tongue, vallecules), locally advanced, rated T3 or T4, whatever the stage N and M0;
* Patient who received curative treatment either surgical (excision and reconstruction free flap) with adjuvant radiotherapy or concurrent chemoradiotherapy;
* Treatment completed at least 12 months prior to study entry;
* Patient whose cancer disease is under control at exam time;
* Subject affiliated to a social security scheme;
* Subject agreeing to participate in the study and who signed the informed consent form.

Exclusion Criteria:

* Minor patient
* No affiliation to a social security scheme (beneficiary or assignee);
* Patient who did not signed the informed consent form
* Patient with neurological disease that can affect the upper airways function
* Patient has already been treated for head and neck cancer;
* Patient has a lesion classified T1 or T2 or M1;
* Patient has received different treatments: surgical resection without reconstruction, only radiotherapy
* Unweaned alcoholic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Measuring the index of apneas and hypopneas (IAH), defined by the number of apneas per sleep hour | 1 day
  For an IAH <10: no Obstructive Sleep Apnea Syndrome (OSAS) For an IAH>30: severe OSAS is diagnosed

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale - Hôpital de la Timone, AP-HM, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided